CLINICAL TRIAL: NCT04228354
Title: A Trial to Demonstrate Bioequivalence Between Semaglutide Drug Product Concentrations 0.68 mg/mL and 1.0 mg/mL
Brief Title: A Research Study Looking at the Comparability (Bioequivalence) of Two Versions of Semaglutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4649; U1111-1241-6257 (Other: World Health Organization (WHO)); 2019-004020-37 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-01-13; First posted 2020-01-14 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide 0.68 mg/mL (Experimental): Semaglutide administered with the PDS290 pen-injector
  Interventions: Drug: Semaglutide
- Semaglutide 1.0 mg/mL (Experimental): Semaglutide administered with the PDS290 pen-injector
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Two doses of semaglutide given by subcutaneous (s.c., under the skin) injection with different drug product concentration and separated by 6 to 8 weeks

SUMMARY:
The study will look at how two different versions of semaglutide reach and stay in the blood after injection. The study aims to show similar levels of semaglutide in the blood when using the different versions. Participants will get both versions of semaglutide. The order in which participants receive the versions is decided by chance. Participants will get the medicines as an injection under the skin of the belly with the use of a pen-injector. The study will last for about 11 to 17 weeks. Participants will have 27 visits with the study doctor. At 2 visits, participants will stay in the clinic for 4 days and 3 nights. Participants may have to stop the study if the study doctor thinks that there are risks for their health. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index between 20.0 and 27.0 kg/m^2 (both inclusive).

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive methods.
* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration curve from 0 to tz | 0-840 hours
  h*nmol/L
Maximum semaglutide plasma concentration | 0-840 hours
  nmol/L

SECONDARY OUTCOMES:
Area under the semaglutide plasma concentration curve | 0-840 hours
  h*nmol/L
Time to Cmax for semaglutide | 0-840 hours
  h
Terminal elimination half-life | 0-840 hours
  h
Total apparent clearance of semaglutide | 0-840 hours
  L/h
Apparent volume of distribution of semaglutide | 0-840 hours
  L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor & Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com